CLINICAL TRIAL: NCT05812625
Title: Effectiveness of Myo-kinetic Stretching Exercises Versus Post-isometrics Relaxation Exercise With Traction in Patients of Cervical Radiculopathy
Brief Title: Myo-kinetic Stretching Versus Post-isometrics Relaxation Exercise With Traction in Patients of Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCRAHS/REC/23/05
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group A (Experimental): • Group A will receive conservative baseline treatment consisted of hot pack therapy for 10 minutes and traction for 8 minutes with Myokinetic stretching technique. Subject will be in supine lying on the plinth and the head will be placed at the edge of the plinth by the therapist. Then with one hand the therapist held the neck in cervical lateral flexion to the opposite side so as to achieve the stretching of the trapezius muscle. Myofascial release by applying sustained finger pressure for 5-10 s on the involved trapezius was given. A gentle myofascial stretching force was applied to take up slack and sustained until a release occurred .The MST protocol comprised of three sets of 4 stretches with 5 seconds rest period between the stretches. Treatment will be provided twice a week for 8 weeks.
  Interventions: Other: Myokinetic stretching technique
- Interventional Group B (Active Comparator): • Group B will be treated by conventional baseline treatment with Post-isometric Relaxation Exercises. Cervical paraspinal post isometric relaxation will be performed with the patient supine, while the therapist will slowly lift the patient's head toward the ceiling. Once a comfortable stretch will be felt, the patient is asked to push their head back (with approximately 10% of their strength), while the therapist will resist the movement; thus, creating an isometric contraction. This position is held for 8-10 seconds. The patient will be asked to inhale deeply and, upon exhalation, will be instructed to relax while the therapist will lift the patient's head a little further towards the ceiling. The protocol will be comprised of three sets of post isometric relaxation with 5 seconds rest period. Treatment will be provided twice a week for 8 weeks.
  Interventions: Other: Post Isometric Relaxation

INTERVENTIONS:
Other: Myokinetic stretching technique — Myokinetic stretching technique (MST) is a form of myofascial release, which involves active or passive stretching and movement as well as muscle energy techniques until a desirable release from the taut band is achieved.
  Arms: Interventional Group A
Other: Post Isometric Relaxation — Post Isometric Relaxation (PIR) is the effect of the decrease in muscle tone in a single or group of muscles, after a brief period of submaximal isometric contraction of the same muscle.
  Arms: Interventional Group B

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of Myo-kinetic stretching exercises versus post-isometric relaxation exercise in patients with cervical radiculopathy. Convenient sampling technique will be used to enroll the patients. Patients will be screened on the basis of pre formulated eligibility criteria. Written Consent will be taken from each patient for participation in the trial. The calculated Sample size of this study will be 68 calculated through Epitool. Group A will receive conservative baseline treatment consisted of hot pack therapy for 10 minutes and traction for 8 minutes. Myo-kinetic stretching exercises and group B will receive conservative baseline treatment and post-isometric relaxation exercise. The assessment of patients will be done at baseline, 4th and 8th week. The outcomes from patients will be calculated by using Numeric Pain Rating Scale (NPRS), Goniometer and Neck Disability Index. The comparison between pre-treatment and post-treatment data will be done after 8th week. Data will be analyzed through SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Duration of cervical pain more than 4 weeks.
* History of positive Spurling test

Exclusion Criteria:

* History of previous cervical surgery
* Cervical spine tumor.
* Rheumatoid arthritis, prolong steroid use and osteoporosis in cervical region.
* Cervical spine fracture.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
Cervical Pain | 8 weeks
  Cervical Pain will be measured by Numeric Pain Rating Scale
Neck Disability | 8 weeks
  Neck disability will be measured by Neck Disability Index
Cervical Range of motion | 8 weeks
  Cervical Range of motion will be measured by Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Sahreen Anwar, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- Allied Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No